CLINICAL TRIAL: NCT02665325
Title: Cognitive Functions and Mood During Thyrotropin Suppressive Therapy in Patients With Differentiated Thyroid Carcinoma
Brief Title: Cognitive Functions During Thyrotropin Suppressive Therapy in Patients With Differentiated Thyroid Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Inner Mongolia Medical University (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Sponsor
Other Study IDs: AHInnerMongolia-Thyroid-01
Record Dates: First submitted 2016-01-17; First posted 2016-01-27 (Estimated); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Cognitive Impairment
Keywords: TSH-suppressive therapy; cognitive function
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Thyroidectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- TSHsuppressive therapy group: TSH-suppressive therapy group: newly diagnosed differentiated thyroid carcinoma and undergone thyroidectomy according to the China thyroid association guidelines for the Management of thyroid nodule and thyroid cancer; followed by TSH-suppressive therapy 6 /12 months.
  Interventions: Drug: TSH-suppressive therapy
- Negative control group: Healthy volunteers (normal T3,T4,FT3,FT4,TSH, TG-ab,TPO-ab,TG) are recruited to match the patients with age, gender, education level, ect.
- Positive control group: Newly diagnosed nodular goiter and undergone thyroidectomy according to the China thyroid association guidelines for the management of thyroid nodule and thyroid cnacer; followed by L-T4 replacement therapy 6/12 months.

INTERVENTIONS:
Drug: TSH-suppressive therapy — Thyroidectomy according to the China thyroid association guidelines for the Management of thyroid nodule and thyroid cancer; followed by TSH-suppressive therapy 6 /12 months.
  Other Names: Thyroidectomy
  Groups: TSHsuppressive therapy group

SUMMARY:
Thyroid carcinoma is the common endocrine system malignant neoplasm. At present it has become the malignant neoplasm of fastest growing incidence rate. More than 90% thyroid carcinoma is thyroid differentiated carcinoma（DTC）. Postoperative oral L-thyroxine suppressing thyroid stimulating hormone (TSH) treatment is the standard therapy in DTC patients. While TSH-suppressive therapy with L-thyroxine can cause subclinical hyperthyroidism in treatment of patients with thyroid differentiated carcinoma. The impact of this therapy on cognitive functions and mood have not been systematically studied. The investigators infer the subclinical hyperthyroidism caused by TSH-suppressive therapy may impact cognitive function and mood disorders in DTC patients. The aim of this study is to explore the possible mechanism of cognitive function impairment in the course of TSH-suppressive therapy by rat model of total thyroidectomy + TSH-suppressive therapy and clinical trials. The result of this study may provide clinical and experimental basis for the side effects risk result form TSH-suppressive therapy in DTC patients.

DETAILED DESCRIPTION:
1. Object:

   Patients aged 18-65 years; newly diagnosed differentiated thyroid carcinoma and undergone thyroidectomy according to the China thyroid association guidelines for the Management of thyroid nodule and thyroid cancer; followed by TSH-suppressive therapy 6 /12 months.
2. Clinical information, examination data and neuropsychological assessments:

Information is obtained from medical record abstraction. Serum T3, T4, FT3, FT4, TSH, TG-ab, TPO-ab, TG levels and neuropsychological assessments are examined after TSH-suppressive therapy 6 /12 months. Cognitive complaints were assessed with the Mini-Mental State Examination (MMSE), Clock Drawing Test (CDT), Digit Symbol test (DST), Wechsler Memory Scale (WMS), Aphasia Battery of Chinese （ABC） and patient health questionnaire-9 (PHQ-9).

Healthy volunteers (normal T3, T4, FT3, FT4, TSH, TG-ab, TPO-ab, TG) are recruited to match the patients with age, gender, education level, etc.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed differentiated thyroid carcinoma.
* Undergo thyroidectomy according to the China thyroid association guidelines for the Management of thyroid nodule and thyroid cancer.
* Followed by TSH-suppressive therapy 6 /12 months.

Exclusion Criteria:

* Current or past disorder/disease of the central nervous system or medical condition impacting cognitive functioning.
* Head trauma history with prolonged loss of consciousness.
* Epilepsy, dementia, or learning disability.
* Current or past psychotic-spectrum disorder or current major affective disorder.
* Current substance abuse/dependence.
* Daily tobacco and alcohol use.
* Whole brain irradiation or surgery.
* Prior cancer diagnosis or chemotherapy treatment.
* Active autoimmune disorder.
* Insulin-dependent diabetes.
* Uncontrolled allergic condition or asthma.
* Chronic use of oral steroid medication.
* Hormone therapy (estrogen, progestin compounds).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-65 years; newly diagnosed differentiated thyroid carcinoma and undergone thyroidectomy according to the China thyroid association guidelines for the Management of thyroid nodule and thyroid cancer; followed by TSH-suppressive therapy 6 /12 months.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-01; Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Cognitive impairment assessed with the Mini-Mental State Examination (MMSE) | 2 years
Cognitive impairment assessed with the Clock Drawing Test (CDT) | 2 years
Cognitive impairment assessed with the Digit Symbol test (DST) | 2 years
Cognitive impairment assessed with the Wechsler Memory Scale (WMS) | 2 years
Cognitive impairment assessed with the Aphasia Battery of Chinese （ABC） | 2 years
Mood assessed with the patient health questionnaire -9 (PHQ-9) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Shan Jin, PhD, Study Director — The Affiliated Hospital of Inner Mongolia Medical University
Locations (1):
- Shan Jin, Hohhot, Inner Mongolia, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fiore E, Vitti P. Serum TSH and risk of papillary thyroid cancer in nodular thyroid disease. J Clin Endocrinol Metab. 2012 Apr;97(4):1134-45. doi: 10.1210/jc.2011-2735. Epub 2012 Jan 25. PMID 22278420
- [Background] Biondi B, Cooper DS. Benefits of thyrotropin suppression versus the risks of adverse effects in differentiated thyroid cancer. Thyroid. 2010 Feb;20(2):135-46. doi: 10.1089/thy.2009.0311. PMID 20151821
- [Background] Davis PJ, Zhou M, Davis FB, Lansing L, Mousa SA, Lin HY. Mini-review: Cell surface receptor for thyroid hormone and nongenomic regulation of ion fluxes in excitable cells. Physiol Behav. 2010 Feb 9;99(2):237-9. doi: 10.1016/j.physbeh.2009.02.015. Epub 2009 Feb 25. PMID 19248795
- [Background] Bauer M, Silverman DH, Schlagenhauf F, London ED, Geist CL, van Herle K, Rasgon N, Martinez D, Miller K, van Herle A, Berman SM, Phelps ME, Whybrow PC. Brain glucose metabolism in hypothyroidism: a positron emission tomography study before and after thyroid hormone replacement therapy. J Clin Endocrinol Metab. 2009 Aug;94(8):2922-9. doi: 10.1210/jc.2008-2235. Epub 2009 May 12. PMID 19435829
- [Background] Puighermanal E, Busquets-Garcia A, Maldonado R, Ozaita A. Cellular and intracellular mechanisms involved in the cognitive impairment of cannabinoids. Philos Trans R Soc Lond B Biol Sci. 2012 Dec 5;367(1607):3254-63. doi: 10.1098/rstb.2011.0384. PMID 23108544
- [Result] Wekking EM, Appelhof BC, Fliers E, Schene AH, Huyser J, Tijssen JG, Wiersinga WM. Cognitive functioning and well-being in euthyroid patients on thyroxine replacement therapy for primary hypothyroidism. Eur J Endocrinol. 2005 Dec;153(6):747-53. doi: 10.1530/eje.1.02025. PMID 16322379